CLINICAL TRIAL: NCT05288309
Title: The Effect Of Use Of Raınstick And Kaleydoscope On Paın Anxıety And Parent Satısfactıon Durıng Blood Draw In Chıldren: A Randomızed Controlled Study
Brief Title: The Effect Of Use Of Raınstick And Kaleydoscope On Paın Anxıety Durıng Blood Draw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Gülsün Ayran, Asistant Professor, Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Erzi̇ncanBYÜ
Record Dates: First submitted 2022-02-03; First posted 2022-03-21 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Pain; Child, Only; Anxiety; Pain, Procedural
Keywords: Anxiety; Blood draw; children; Nursing; Pain; Rainstick; Kaleidoscope
MeSH Terms: conditions — Pain; Anxiety Disorders; Pain, Procedural

STUDY DESIGN:
Who Masked: Participant
Masking Description: Children in the 5-12 age group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAİNSTİCK (Other): In the 1st experimental group, the sound of the rain stick was played to distract attention. The rainstick, used by traditional societies, is a rhythm instrument that makes the sound of rain by moving it up and down. The length of the rain stick made of bamboo is 40 cm. There are spiral-shaped spines inside the tool, which is closed at both ends. It makes the sound of drizzling rain by moving it up and down.
  Interventions: Other: RAINSTİCK
- KALEİDOSCOPE (Other): In the second experimental group, kaleidoscope was used to distract attention. A kaleidoscope, or kaleidoscope, is a device that sees colorful patterns when looked into. Inside, there are three mirrors adjacent to each other with an inclination of 60 degrees between them. There are pieces of colored glass between the mirrors. When viewed from one end of this binocular, shape-shifting polygons are seen, often with images that will never be the same again. These patterns are created by the reflection of light and change constantly as the binoculars are moved.
  Interventions: Other: KALEİDOSCOPE

INTERVENTIONS:
Other: RAINSTİCK — When the child, who was taken to Experimental Group 1, sat on the patient's chair, the sound of the rain stick was started to be played 1 minute before the blood draw. At that time, the nurse began to prepare the child for the blood draw. The tourniquet insertion procedure and the determination of the vein from which blood will be drawn from the antecubital region were performed by the nurse. Blood collection was taken from the antecubital region in one go by the same nurse by means of a vacuum blood collection tube, and blood flowed to the vacuum within 5 seconds, showing that the procedure was successful. This process took about 2-3 minutes and the children listened to the sound of rain sticks throughout the process.
  Arms: RAİNSTİCK
Other: KALEİDOSCOPE — The child, who was taken into Experimental Group 2, was started to watch the kaleidoscope 1 minute before the blood draw, as he sat on the patient's chair. At that time, the nurse began to prepare the child for the blood draw. The tourniquet insertion procedure and the determination of the vein from which blood will be drawn from the antecubital region were performed by the nurse. Blood collection was taken from the antecubital region in one go by the same nurse by means of a vacuum blood collection tube, and blood flow to the vacuum within 5 seconds showed that the procedure was successful. This process took about 2-3 minutes and children were watched with kaleidoscope throughout the process.
  Arms: KALEİDOSCOPE

SUMMARY:
Medical procedures are negative experiences that cause pain, distress, and anxiety and are not only uncomfortable during medical procedures, especially in children; negative consequences such as poor recovery, sleep disturbances, and post-traumatic stress symptoms. There are many different approaches, including pharmacological and non-pharmacological methods, for the treatment of pain and anxiety in children during medical procedures. Non-pharmacological methods vary depending on the child's age, level of development and the type of procedure, and non-pharmacological methods generally used in children fall into three groups: supportive, physical and cognitive or behavioral methods. Supportive methods are practices that include psychosocial care of the child, such as reading a book or playing games. Physical methods include techniques such as cold application, massage, and transcutaneous electrical nerve stimulation. Cognitive or behavioral methods include practices such as listening to music, daydreaming, relaxation, and various methods of distraction. Cognitive and behavioral approaches typically use the activating or relaxing effects of music for arousal or calming and to enhance the learning of certain skills and behaviors. Music therapy practice reduces pain and anxiety levels by stimulating the pituitary gland.

Another method used is the use of kaleidoscope. In the literature, they reported that the use of kaleidoscope is effective in reducing the pain that may occur during blood collection in studies conducted with preschool and school children, children and adolescents, and school-age children. The results show that the kaleidoscope can be used effectively to distract children from the painful procedure and reduce the perception of pain.

DETAILED DESCRIPTION:
Data Collection After obtaining the necessary institutional permissions, parents and children will be informed about the research through the "Informed Voluntary Consent Form" in the interview room 15 minutes before the blood draw. Research data will be collected by the researcher by face-to-face interview technique. A questionnaire including questions such as the age of the child, the time of the last blood draw, the parent's presence with the child will be applied to the parents. To ensure randomisation, children will be asked to choose one of the sealed envelopes. Then, the blood collection room will be passed to perform the procedure.

When the child to be taken to Experimental Group 1 sits in the patient's chair, the sound of the rain stick will be played 1 minute before the blood draw. The nurse will then begin to prepare the child for the blood draw. The tourniquet insertion procedure and the determination of the vein from which blood will be drawn from the antecubital region will be performed by the nurse. Blood collection will be taken from the antecubital region at once by the same nurse through the vacuum blood collection tube, and blood flow to the vacuum within 5 seconds will show that the procedure is successful. In the meantime, a pulse oximeter will be attached to the index finger of the hand on the other arm, where blood is not drawn, and the heart rate will be evaluated before the procedure and after the procedure. This process will take about 2-3 minutes and the children will listen to the sound of the rain stick throughout the process. After the procedure is over, the children will be taken out of the blood collection room and taken to the waiting area, and they will be asked to determine the severity of pain they feel during the procedure. WBFPS will be used to find out how much pain the child has during the blood draw, and ÇAS-D will be used to determine the anxiety state. Pain and anxiety level will be evaluated by the child, nurse, parent and researcher.

The Kaleidoscope will start to be watched 1 minute before the blood draw process, as the child, who will be taken into Experimental Group 2, sits in the patient's chair. The nurse will then begin to prepare the child for the blood draw. The tourniquet insertion procedure and the determination of the vein from which blood will be drawn from the antecubital region will be performed by the nurse. Blood collection will be taken from the antecubital region at once by the same nurse through the vacuum blood collection tube, and blood flow to the vacuum within 5 seconds will show that the procedure is successful. In the meantime, a pulse oximeter will be attached to the index finger of the hand on the other arm, where blood is not drawn, and the heart rate will be evaluated before the procedure and after the procedure. This process will take about 2-3 minutes, and children will be shown a kaleidoscope image throughout the process. After the procedure is over, the children will be taken out of the blood collection room and taken to the waiting area, and they will be asked to determine the severity of pain they feel during the procedure. WBFPS will be used to find out how much pain the child has during the blood draw, and ÇAS-D will be used to determine the anxiety state. Pain and anxiety level will be evaluated by the child, nurse, parent and researcher.

No interventional procedure will be applied to the children in the control group. The blood collection will be arranged in such a way that it is taken from the antecubital region in one go by the same nurse by means of a vacutainer. In the meantime, a pulse oximeter will be attached to the index finger of the hand on the other arm, where blood is not drawn, and the heart rate will be evaluated before the procedure and after the procedure. After the procedure is over, the children will be taken out of the blood collection room and taken to the waiting area. WBFPS will be used to find out how much pain the child has during the blood draw, and ÇAS-D will be used to determine the anxiety state. Pain and anxiety level will be evaluated by the child, nurse, parent and researcher. In both groups, parents will be provided with their children in the blood collection room during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 5-12 years old
* There should be no pain before the blood draw procedure
* Should not have a chronic disease that will cause pain Blood should be taken from the antecubital region
* Must be willing to participate in the research

Exclusion Criteria:

* The transmission barrier
* Wearing glasses
* Involuntary

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Comparison of Wong-Baker Faces Pain Scale Mean Scores by Groups | It will be evaluated within an average of 5 minutes during the blood collection process.
  This scale measuring the severity of pain was used in children aged between 3-18 years. In this scale, pain was scored for facial expressions according to numerical values, and the numerical rating of the scale varied between 0 and 10. Facial expressions ranging from smiling (0=very happy/no pain) to crying (10=most painful) indicated emotions.

SECONDARY OUTCOMES:
Comparison of Child Anxiety Scale Mean Scores before and during the procedure according to the groups | It will be evaluated within an average of 3 minutes before the blood draw and an average of 3 minutes during the blood collection process.
  CSAS was a thermometer-like scale with a light bulb at the bottom and horizontal upward lines at intervals. On the scale, the children were instructed as "Imagine all your anxious or frustrated feelings are in the bulb or bottom of the thermometer." "If you're a little worried or nervous, emotions can go a little upward on the thermometer. If you are very, very anxious or nervous, the emotions can go to the top. Put a line indicating how worried or angry you are on the thermometer." A transparent meter with increments of ½ point marked was placed above the rating of children, then the increment of ½ point was rounded to the nearest number. The score varied between 0 and 10

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Erzincan Binali Yıldırım University, Merkez, Erzi̇ncan
  - Erzincan Binali Yıldırım Üniversitesi, Merkez, Erzi̇ncan